CLINICAL TRIAL: NCT02343653
Title: The Effect of Resistance Training on Muscle Strength and Nutritional Status in Patients With Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Training/Cirrhosis
Record Dates: First submitted 2015-01-09; First posted 2015-01-22 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Liver Cirrhosis
Keywords: Malnutrition; Muscle mass; Nutrition
MeSH Terms: conditions — Liver Cirrhosis; Malnutrition | interventions — Nutritional Status; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition (Active Comparator): Participants receive a controlled diet consisting of 1.2-1.5 g of protein/kg/day for 12 weeks according to guidelines for enteral nutrition and patients with cirrhosis. The group receives dietary guidance and protein supplements.
  Interventions: Behavioral: Nutrition
- Nutrition and strength training (Experimental): Participants in this group receive same controlled diet consisting of 1.2-1.5 g of protein/kg/day for 12 weeks as the "No intervention"-group. Participants will also receive supervised strength training 3 x 60 min./week for 12 weeks. The group receives dietary guidance and protein supplements, which on training days should be consumed within 30 minutes after exercise.
  Interventions: Behavioral: Nutrition and strength training

INTERVENTIONS:
Behavioral: Nutrition and strength training — All participants will receive professional dietary guidance and a protein supplement. At the beginning and end of the intervention every participant will be part of a program consisting of:
  Test of muscle strength, blood samples, assessment of nutritional status, MRi scan, test of Quality of life by questionnaire and test of the ammonium metabolism. After one year readmissions will by registered.
  The intervention group will receive supervised training.
  Arms: Nutrition and strength training
Behavioral: Nutrition — All participants will receive professional dietary guidance and a protein supplement. At the beginning and end of the intervention every participant will be part of a program consisting of:
  Test of muscle strength, blood samples, assessment of nutritional status, MRi scan, test of Quality of life by questionnaire and test of the ammonium metabolism. After one year readmissions will by registered.
  Arms: Nutrition

SUMMARY:
The purpose is to investigate the effect of strength training on muscle strength, muscle mass and nutritional status in patients with liver cirrhosis to clarify possible metabolic and inflammatory changes during this intervention. In addition the investigator examine if the intervention is associated with fewer hospital readmission and an improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis, Child Pugh score A and B

Exclusion Criteria:

* Cirrhosis, Child-Pugh score C at inclusion
* Neurological and/or psychiatric disorder
* Pregnancy, breastfeeding
* Patients with malignancy
* Patients with hepatic encephalopathy at inclusion
* Patients with atypical diets, such as vegans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Maximal voluntary muscle strength in knee extensor will be measured by an isokinetic dynamometer and hand strength by hand dynamometer. | 12-14 weeks

SECONDARY OUTCOMES:
Nutritional status as measured by Triceps skinfold thickness (TSF), mid-upper-arm circumference (MUAC), mid-arm muscle area (MAMA) and hand dynamometer | 12-14 weeks
Readmissions as measured by a follow-up one year after the intervention. | 1-1,5 year
Quality of Life as measured by a standardized questionnaire (SF-36) | 12-14 weeks
Insulin sensitivity as measured by HOMA-IR | 12-14 weeks
Ammonia metabolism as measured by Oral Glutamine Challenge Test | 12-14 weeks
  Minimal risk in the taking of blood samples. The participant can experience nausea and dizziness but will not be left unsupervised during the test.
Muscle mass as measured by MRi scan and bioimpedance scan. | 12-14weeks

CONTACTS AND LOCATIONS:
Overall Officials: Niels Kristian Aagaard, Chief phys., Study Director — Department of Hepatology and Gastroenterology V, Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology V, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Aamann L, Dam G, Borre M, Drljevic-Nielsen A, Overgaard K, Andersen H, Vilstrup H, Aagaard NK. Resistance Training Increases Muscle Strength and Muscle Size in Patients With Liver Cirrhosis. Clin Gastroenterol Hepatol. 2020 May;18(5):1179-1187.e6. doi: 10.1016/j.cgh.2019.07.058. Epub 2019 Aug 5. PMID 31394282